CLINICAL TRIAL: NCT00564629
Title: A Phase III, Randomized, Double-Blind, Double-Dummy, Single-Dose Study of the Efficacy and Safety of Intravenous Acetaminophen Versus Oral Acetaminophen for the Treatment of Endotoxin-Induced Fever in Healthy Adult Males
Brief Title: Study of the Efficacy and Safety of Intravenous vs Oral Acetaminophen for Treatment of Fever in Healthy Adult Males
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPI-APF-303
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Fever
MeSH Terms: conditions — Fever | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV acetaminophen plus oral placebo. (Experimental): Administration of a 1 ng/kg body weight test dose of RSE to test for fever response. Observation period of at least 60 minutes to ensure no exaggerated systemic responses, followed by administration of a 4 ng/kg of RSE to induce fever. Randomization to receive 1 g of acetaminophen in 100 ml of intravenous solution and oral placebo.
  Interventions: Drug: Intravenous acetaminophen plus oral placebo; Biological: Reference standard endotoxin (RSE)
- Oral acetaminophen plus IV placebo. (Active Comparator): Administration of a 1 ng/kg body weight test dose of RSE to test for fever response. Observation period of at least 60 minutes to ensure no exaggerated systemic responses, followed by administration of a 4 ng/kg of RSE to induce fever. Randomization to receive oral acetaminophen 1 g plus 100 ml of intravenous placebo solution.
  Interventions: Drug: Oral acetaminophen plus IV placebo; Biological: Reference standard endotoxin (RSE)

INTERVENTIONS:
Drug: Intravenous acetaminophen plus oral placebo — Single dose of 1 gm IV acetaminophen
  Other Names: IV APAP
  Arms: IV acetaminophen plus oral placebo.
Drug: Oral acetaminophen plus IV placebo — Single dose of 1 g PO APAP
  Other Names: IV APAP
  Arms: Oral acetaminophen plus IV placebo.
Biological: Reference standard endotoxin (RSE) — To subjects in both study arms: Administration of a 1 ng/kg body weight test dose of RSE to induce fever and test for fever response. Observation period of at least 60 minutes to ensure no exaggerated systemic responses, followed by administration of a 4 ng/kg of RSE to induce fever.
  Other Names: RSE

SUMMARY:
To assess the rapidity of onset of antipyretic effect and the efficacy and safety of a single dose of IV acetaminophen (IV APAP) versus oral (PO) acetaminophen in the treatment of fever induced by a standard dose of endotoxin

DETAILED DESCRIPTION:
A Phase III, Randomized, Double-Blind, Double-Dummy, Single-Dose Study of the Efficacy and Safety of Intravenous Acetaminophen Versus Oral Acetaminophen for the Treatment of Endotoxin-Induced Fever in Healthy Adult Males

ELIGIBILITY:
Inclusion Criteria (Screening) To be eligible for entry into the Study, Subjects must meet all of the following criteria at Screening:

* Provide written Informed Consent prior to participation in the Study
* Be a healthy male between the ages of 18 and 75 years of age, inclusive, at Randomization
* Have a Body Mass Index (BMI) ≥ 19 and ≤ 45 lbs/in2
* Have the ability to read and understand the Study procedures and have the ability to communicate meaningfully with the Study Investigator and staff
* Be free of physical, mental, or medical conditions which, in the opinion of the Investigator, may confound quantifying assessments for the Study
* Be willing to abstain from smoking cigarettes or using nicotine products from the time of admission to Clinic until Study Completion

Inclusion Criteria (Pre-Randomization) To be eligible for Randomization, Subjects must meet each of the following criteria:

* Be free of evidence of infection based upon clinical assessment and blood (Complete Blood Count- CBC) and urine testing
* Have an average baseline oral temperature that is equal to or below 37 ºC (98.6 ºF) and does not vary more than 0.4 ºC (0.7 ºF) from lowest to highest on three assessments performed during a 30-minute period
* Not develop a medically significant allergic or exaggerated systemic response to administration of a test dose of reference standard endotoxin
* Develop a core temperature of at least 38.6 ºC (101.5 ºF) after IV reference standard endotoxin dosed per Study guidelines and have a fever response to endotoxin that is at or near the peak temperature by virtue of two consecutive temperature assessments 5 minutes apart that are within 0.2 ºC (0.4 ºF) of each other

Exclusion Criteria:

* Has been treated with any medication having antipyretic effects (e.g., corticosteroid,non-steroidal anti-inflammatory drug [NSAID], aspirin, or acetaminophen) within 2 days of clinic admission (aspirin at low dose for cardiac prophylaxis is allowed, but should not be taken on the day of the Study)
* Has significant medical disease(s), laboratory abnormalities, or condition(s) that in the Investigator's judgment could compromise the Subject's welfare, ability to communicate with the Study staff, complete Study activities, or would otherwise contraindicate Study participation
* Has known hypersensitivity or contraindication to receiving endotoxin that in the Investigator's clinical judgment merits discontinuation from further Study participation
* Has known hypersensitivity to acetaminophen, the inactive ingredients (excipients) of the intravenous (IV) or oral (PO) acetaminophen formulation or the Rescue Medications (ibuprofen, aspirin, and ketorolac)
* Has known or suspected recent history of alcohol or drug abuse or dependence as defined by Diagnostic Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria
* Has a history of nasal polyps, angioedema, significant or actively treated bronchospastic disease, or any other significant medical condition that contraindicates participation in the Study or receiving endotoxin, Study Medication, or Rescue Medication
* Has an active infection or other disease or condition that may cause abnormal alterations in body temperature
* Has impaired liver function, e.g.Alanine aminotransferase (ALT) greater than or equal to 3 times the upper limit of normal, bilirubin greater than 3.0, active hepatic disease, or evidence of clinically significant liver disease (e.g., cirrhosis or hepatitis)
* Has participated in another clinical Study (investigational or marketed product) within 30 days of Screening

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New Orleans Center for Clinical Research-Knoxville, Knoxville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy Adult males at one site in the United States
Pre-assignment Details: Eligible subjects were given intravenous (IV) endotoxin 1 ng/kg as a test dose and observed for 1 hour. Next, subjects were administered a 4 ng/kg pyrogenic IV endotoxin dose and monitored until a core temperature of at least 38.6 ºC was reached. Subjects achieving a sufficient fever response were then randomly assigned to study treatments.
Groups:
- Oral Acetaminophen (PO APAP) 1 g: group of subjects randomly selected to receive 1 g of oral acetaminophen as the study treatment
- Intravenous Acetaminophen (IV APAP) 1 g / 100 ml Solution: group of subjects randomly selected to receive 1 g /100 ml of intravenous acetaminophen solution as the study treatment
Period: Overall Study
Arm/Group | Oral Acetaminophen (PO APAP) 1 g | Intravenous Acetaminophen (IV APAP) 1 g / 100 ml Solution
Started | 51 | 54
Completed | 36 | 45
Not Completed | 15 | 9
Not completed — Vomited within 2 hours of receiving drug | 15 | 9

BASELINE CHARACTERISTICS:
Groups:
- PO APAP 1 g: group of subjects randomly selected to receive 1 g of oral acetaminophen and 100 ml of intravenous placebo solution as the study treatment
- IV APAP 1 g / 100 ml Solution: group of subjects randomly selected to receive 1 g of acetaminophen in 100 ml of intravenous solution and oral placebo as the study treatment
- Total: Total of all reporting groups
Arm/Group | PO APAP 1 g | IV APAP 1 g / 100 ml Solution | Total
Number analyzed (Participants) | 51 | 54 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 54 | 105
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — mITT(modified intent to treat) population was used for age continuous baseline measure. mITT is defined as the all randomized subjects who received at least one full dose of oral or intravenous study medication without vomiting less than 2 hours after the oral study medication dose.
  81 subjects were included in the mITT group with 36 subjects in the oral acetaminophen arm and 45 subjects in the IV acetaminophen arm.
  years | 32.1 (9.07) | 33.8 (11.6) | 33 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 51 | 54 | 105
Region of Enrollment [Number; unit: participants]
  United States | 51 | 54 | 105

OUTCOME MEASURES:

1. Primary Outcome: The Rapidity of Onset of Antipyretic Effect at 2 Hours (Measured as Weighted Sum of Temperature Differences Over 2 Hours, WSTD2)
Description: This outcome measures when the antipyretic effect begins by statistical analysis of WSTD2, which is the weighted sum of temperature differences from the subject's core temperature at each assessment time point through the first 2 hours compared with the subject's core temperature at T0, weighted by the time elapsed between each 2 consecutive time points. The subject's core temperature was measured using an ingestible temperature monitoring capsule and associated data recorder.
Time Frame: 0-2 hours
Population: mITT population defined as all randomized subjects who received at least 1 full dose of oral study medication (subject not vomiting within 2 hours after oral study drug) or 1 full dose of IV study medication(subject having received all 100 mls solution). This analysis was performed with imputation for non-physiological temperature swing zone effect
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Groups:
- IV APAP 1 g / 100 ml Solution: mITT-Intravenous Acetaminophen 1g
- PO APAP 1 g: mITT-Oral Acetaminophen 1 g
Arm/Group | IV APAP 1 g / 100 ml Solution | PO APAP 1 g
Number analyzed (Participants) | 45 | 36
Degrees Celsius | 0.3 (0.41) | 0.6 (0.55)

2. Secondary Outcome: Time to a Reduction in Temperature From T0 to T360 Minutes.
Description: This outcome measures how much time it took to observe a decrease in subjects' core body temperature by 0.8 ºC, 1.0 ºC, and 1.5 ºC from the temperature at T0 and from the temperature at the peak after T0 through T360 (6 hours). The subject's core temperature was measured using an ingestible temperature monitoring capsule and associated data recorder.
Time Frame: 6 hours
Population: Analysis was performed on the mITT population.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IV APAP 1 g / 100 ml Solution | PO APAP 1 g
Number analyzed (Participants) | 45 | 36
Hours
  reduction in temperature of 0.8 ºC from T0 temp | 4.8 (0.96) | 4.7 (1.41)
  reduction in temp of 0.8 ºC from the peak T0-T360 | 3.5 (1.23) | 2.4 (1.16)
  reduction in temperature of 1.0 ºC from T0 temp | 5.1 (0.85) | 5.0 (1.24)
  reduction in temp of 1.0 ºC from the peak T0-T360 | 3.8 (0.87) | 2.9 (1.16)
  reduction in temperature of 1.5 ºC from T0 temp | 5.7 (0.45) | 5.6 (0.64)
  reduction in temp of 1.5 ºC from the peak T0-T360 | 5.1 (0.17) | 4.2 (1.19)

3. Secondary Outcome: Maximum Temperature Reduction Observed From T0 to T360 Minutes
Description: This outcome measures the maximum core temperature reduction observed from T0 to T360 minutes. The subject's core temperature was measured using an ingestible temperature monitoring capsule and associated data recorder.
Time Frame: T0-T360 minutes
Population: Analysis performed on the mITT population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | IV APAP 1 g / 100 ml Solution | PO APAP 1 g
Number analyzed (Participants) | 45 | 36
Degrees Celsius | -0.8 (0.46) | -1.1 (0.42)

4. Secondary Outcome: Subject's Global Evaluation of Study Medication at T360 Minutes
Description: This outcome measures how satisfied the subject was with the study treatment. The subject was asked to answer "Overall, how would you rate study treatments?" at T360 minutes using a 4-point categorical scale (0=poor, 1=fair, 2=good, 3=excellent).
Time Frame: T360 minutes
Population: Analysis performed on the mITT population.
Measure: Number; unit: participants
Arm/Group | IV APAP 1 g / 100 ml Solution | PO APAP 1 g
Number analyzed (Participants) | 45 | 36
participants
  Poor (0) | 0 | 2
  Fair (1) | 7 | 2
  Good (2) | 18 | 11
  Excellent (3) | 20 | 21

5. Secondary Outcome: The Percentage of Subjects With Temperature < 38 ºC and < 38.5 ºC at Any Timepoint During the Time From T0 to T360 Minutes
Description: This outcome measures what percentage of total subjects had a temperature < 38 ºC and < 38.5 ºC at any timepoint during the time from T0 to T360 minutes.
Time Frame: T0 to T360 minutes
Population: Analysis performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | IV APAP 1 g / 100 ml Solution | PO APAP 1 g
Number analyzed (Participants) | 45 | 36
percentage of participants
  temperature < 38 ºC | 40 | 67
  temperature < 38.5 ºC | 84 | 92

6. Secondary Outcome: WSTD3
Description: This outcome measure is a statistical analysis of WSTD3, which is the weighted sum of temperature differences from the subject's core temperature at each assessment time point through the first 3 hours compared with the subject's core temperature at T0, weighted by the time elapsed between each 2 consecutive time points. The subject's core temperature was measured using an ingestible temperature monitoring capsule and associated data recorder.
Time Frame: 0-3 hours
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | IV APAP 1 g / 100 ml Solution | PO APAP 1 g
Number analyzed (Participants) | 45 | 36
degrees Celsius | 0.2 (0.73) | 0.5 (0.85)

7. Secondary Outcome: WSTD4
Description: This outcome measure is a statistical analysis of WSTD4, which is the weighted sum of temperature differences from the subject's core temperature at each assessment time point through the first 4 hours compared with the subject's core temperature at T0, weighted by the time elapsed between each 2 consecutive time points. The subject's core temperature was measured using an ingestible temperature monitoring capsule and associated data recorder.
Time Frame: 0-4 hours
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | IV APAP 1 g / 100 ml Solution | PO APAP 1 g
Number analyzed (Participants) | 45 | 36
degrees Celsius | -0.20 (1.06) | -0.02 (1.12)

8. Secondary Outcome: WSTD5
Description: This outcome measure is a statistical analysis of WSTD5, which is the weighted sum of temperature differences from the subject's core temperature at each assessment time point through the first 5 hours compared with the subject's core temperature at T0, weighted by the time elapsed between each 2 consecutive time points. The subject's core temperature was measured using an ingestible temperature monitoring capsule and associated data recorder.
Time Frame: 0-5 hours
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | IV APAP 1 g / 100 ml Solution | PO APAP 1 g
Number analyzed (Participants) | 45 | 36
degrees Celsius | -0.7 (1.43) | -0.7 (1.41)

9. Secondary Outcome: WSTD6
Description: This outcome measure is a statistical analysis of WSTD6, which is the weighted sum of temperature differences from the subject's core temperature at each assessment time point through the first 6 hours compared with the subject's core temperature at T0, weighted by the time elapsed between each 2 consecutive time points. The subject's core temperature was measured using an ingestible temperature monitoring capsule and associated data recorder.
Time Frame: 0-6 hours
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | IV APAP 1 g / 100 ml Solution | PO APAP 1 g
Number analyzed (Participants) | 45 | 36
degrees Celsius | -1.4 (1.88) | -1.7 (1.70)

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events(TEAEs)were reported from T0 (on or after the start of study medication) to 6 hours after study medication was administered to the subject.
Description: TEAEs are adverse events that start on or after the start of study medication.
Arm/Group | Oral Acetaminophen (PO APAP) 1 g | Intravenous Acetaminophen (IV APAP) 1 g / 100 ml Solution
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/54
Other Adverse Events (participants affected / at risk) | 17/51 | 13/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Acetaminophen (PO APAP) 1 g (N=51) | Intravenous Acetaminophen (IV APAP) 1 g / 100 ml Solution (N=54)
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 13 | 6
Headache (Nervous system disorders) | 4 | 5

LIMITATIONS AND CAVEATS:
Protocol and statistical analysis plan were amended to clarify endpoints prior to database lock and analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the Institution nor the Investigator shall have the right to publish the Institution findings without prior written consent of Cadence.